CLINICAL TRIAL: NCT05606185
Title: Amount of Root Resorption of Maxillary Anteriors After en Masse Versus Two Step Space Closure Using Cone Beam Computed Tomography
Brief Title: Amount of Root Resorption of Maxillary Anteriors After en Masse Versus Two Step Space Closure
Acronym: CBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hiba Tabassum, Dr, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DUHS/BASR/2019/-509
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Root Resorption
Keywords: Two step retraction; En masse retraction; Cone Beam Computed Tomography
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two step retraction (Active Comparator): teeth will be retracted in two stages
  Interventions: Procedure: retraction method
- En masse retraction (Experimental): teeth will be retracted in one stage
  Interventions: Procedure: retraction method

INTERVENTIONS:
Procedure: retraction method — Three dimensional evaluation of root resorption using cone beam computed tomography

SUMMARY:
The goal of this study is to compare the three dimensional root resorption after extraction space closure in two groups: two step retraction and en masse retraction. Th main aim of this study is to conclude which method is less damaging to the roots.

Participants will be divided into two groups:

1. En masse retraction (experimental)
2. Two step retraction (control) Pre retraction and post retraction CBCT scans will be compared for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent to be part of this study.
* Patients with Class I or Class II malocclusion.
* Patients requiring extractions of maxillary first premolars with absolute anchorage.
* Good periodontal status.

Exclusion Criteria:

* Patients who are syndromic or have cleft lip and/or palate.
* Patients with severe root dilacerations or root canal treated incisors.
* Patients receiving drugs that alter tooth movement.
* Patients with systemic disease like endocrinological disorders, vit D excess or deficiency, thyroid or parathyroid problems.
* Patients with history of trauma to dentition or impacted teeth in anterior maxilla.
* Patients who have undergone previous orthodontic treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Root resorption | 8 months
  Amount of root resorption in three dimensions

CONTACTS AND LOCATIONS:
Overall Officials: HIBA Tabassum, MDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No